CLINICAL TRIAL: NCT05414773
Title: Zeiss® IOLMaster 700 Corneal Topography Module Comparison With Schwind's Sirius Corneal Topography®
Acronym: VIMECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Edouard KOCH (Other)
Responsible Party: Sponsor-Investigator, Edouard KOCH, Investigator Coordinator, Versailles Hospital
Organization: Versailles Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P21/19
Record Dates: First submitted 2022-06-03; First posted 2022-06-10 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corneal Topography with IOLMaster and Sirius topography. (Experimental): The experimental group will have the two exams: the topography with the IOLMAster and the topography with Sirius topography.
  Interventions: Other: measurement of axial length and keratometry by sonographers with a topographic module

INTERVENTIONS:
Other: measurement of axial length and keratometry by sonographers with a topographic module — measurement of axial length and keratometry by sonographers with a topographic module

SUMMARY:
In order to determine the intraocular lens to be implanted during cataract surgery, keratometry and axial length must be measured in preoperative. The axial length is obtained by ocular ultrasound mode B. Keratometry is obtained by means of an automatic refractometer or corneal topography. Currently, ultrasound scanners are being developed with a topography module to combine axial length and keratometry measurement. The investigators want to evaluate the corneal topography module of the Zeiss® IOL Master 700 biometer.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women Requiring CHV Cataract Surgery
* Aged 18 or over
* Insured under a social security scheme
* Having been informed of the clinical study and having given oral express consent

Exclusion Criteria:

* Person unable to express consent
* Patient with a history of corneal dystrophy, corneal refractive surgery or keratoconus.
* History of chronic corneal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
keratometry measurements | day 1
  to show that the keratometry measurements obtained using the topography module integrated in the IOL Master 700 are consistent with those obtained by a standard topography in patients operated for cataract surgery. The measures will be: K1 (steepest corneal meridian), K2 (flattest corneal meridian), Kmax (central corneal keratometry), the unit of measurement is the diopter.

IPD SHARING:
Plan to Share IPD: Undecided